CLINICAL TRIAL: NCT03832985
Title: Reporting Adult-Onset Genomic Results to Pediatric Biobank Participants and Parents
Brief Title: Pediatric Reporting of Adult-Onset Genomic Results
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Adam Buchanan, Associate Professor and Chair, Geisinger Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0419; 1R01HG009671-01A1 (NIH)
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome; Lynch Syndrome; Familial Hypercholesterolemia
Keywords: adult-onset; pediatric; genomic; genetic
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: The study sample will be drawn from all pediatric MyCode participants (ages 0-17 years). At least one parent will be enrolled for each pediatric participant. Parents of children ages 0-10 years at enrollment will participate in data collection; parents of children ages 11-17 years at enrollment and their children will participate in data collection. Group 3 participants will be frequency matched to Groups 1 and 2 participants on age and sex.
  Individuals who have already had genetic counseling for any of the MyCode target conditions as part of their routine clinical care will be excluded to avoid confounding study findings.
  Quantitative data collection will be on 705 (530 parents and 175 adolescents).
Masking Description: No one is prevented from having knowledge of this project.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Receive an adult-onset result (Experimental): Compare change in psychosocial outcomes and health behaviors of those with a pathogenic variant in a gene associated with adult onset of disease.
  Interventions: Genetic: Receive an adult-onset result
- Receive a pediatric-onset result (Experimental): Compare change in psychosocial outcomes and health behaviors of those with a pathogenic variant in a gene associated with pediatric onset of disease or with risk reduction interventions that begin in childhood.
  Interventions: Genetic: Receive a pediatric-onset result
- Control - No result (Active Comparator): Compare change in psychosocial outcomes and health behaviors of those without a genomic result.
  Interventions: Genetic: Control - No Result

INTERVENTIONS:
Genetic: Receive an adult-onset result — Assess the psychosocial outcomes and the lived experience of MyCode pediatric participants and parents who have received an adult-onset genomic result.
  Arms: Receive an adult-onset result
Genetic: Receive a pediatric-onset result — Assess the psychosocial outcomes and the lived experience of MyCode pediatric participants and parents who have received an adult-onset genomic result.
  Arms: Receive a pediatric-onset result
Genetic: Control - No Result — Assess the psychosocial outcomes and the lived experience of MyCode pediatric participants and parents who have not received an adult-onset genomic result.
  Arms: Control - No result

SUMMARY:
The Investigators will conduct a longitudinal, mixed-methods cohort study to assess primary and secondary psychosocial outcomes among 705 MyCode pediatric participants and their parents, and health behaviors of parents whose children receive an adult- or pediatric-onset genomic result. Data will be gathered via quantitative surveys using validated measures of distress, family functioning, quality of life, body image, perceived cancer/heart disease risk, genetic counseling satisfaction, genomics knowledge, and adjustment to genetic information; qualitative interviews with adolescents and parents; and electronic health records review of parents' cascade testing uptake and initiation of risk reduction behaviors. The investigators will also conduct empirical and theoretical legal research to examine the loss of chance doctrine and its applicability to genomic research.

DETAILED DESCRIPTION:
The Investigators propose a longitudinal, observational cohort study using mixed methods to compare change in psychosocial outcomes and health behaviors among three study groups of pediatric MyCode participants and their parents:

1. Group 1 - those with a pathogenic variant in a gene associated with adult onset of disease (n=17 adolescents, 50 parents)
2. Group 2 - those with a pathogenic variant in a gene associated with pediatric onset of disease or with risk reduction interventions that begin in childhood (n=53 adolescents, 160 parents)
3. Group 3 - those who do not receive a genomic result (n=105 adolescents, 320 parents)

The Investigators will use the current existing MyCode list of actionable genes designated as actionable by the American College of Medical Genetics and Genomics. Parents of pediatric MyCode participants will be offered the opportunity to participate in the study prior to learning to which group they belong. Consistent with Geisinger policy, children ages 7-17 will be asked to give assent to participate. If a child does not want to assent to participate, he or she will not be enrolled into the study (regardless of their parents' preference regarding enrollment). Parents of children who do not give assent will be ineligible to participate. Parents who decline participation when their child is suspected to have a pathogenic adult-onset result will have their child's sample held for clinical confirmation until the child reaches age 18 years. Parents who decline participation when their child is suspected to have a pathogenic pediatric-onset result will proceed to clinical confirmation of the result and, if confirmed, follow the established clinical return procedure. This recruitment approach is consistent with the MyCode philosophy of notifying participants of actionable findings. Parent-participants will be asked to assess psychosocial outcomes for themselves and for their children. Consistent with co-investigator Angela Bradbury's research on the experience of adolescent girls from families at increased risk for breast cancer, pediatric participants ages 11-17 years at enrollment (i.e., adolescents) will also participate in quantitative surveys and qualitative interviews.

Psychosocial variables such as anxiety and depression will be assessed among parents and adolescents at enrollment (T1), after which those suspected of having a pathogenic variant will proceed to clinical confirmation of that variant. Those whose variant is confirmed clinically as pathogenic or likely pathogenic will then be scheduled for a disclosure appointment. These appointments will be conducted by a genetic counselor and psychologist, who will perform psychosocial assessment, conduct therapeutic consults as needed, and conduct periodic psychosocial assessments of adolescent participants with adult-onset results. Participants with suspected pathogenic variants that are not confirmed clinically and participants without a suspected pathogenic variant will be scheduled for a study visit to notify them of their group status and remind them to follow up with their pediatrician if they have significant personal or family history of cancer or heart disease.

Validated surveys will be used to measure outcomes in each study group at 1 month (T3), 6 months (T4) and 12 months (T5) post-disclosure visit. The investigators will conduct qualitative interviews with a subset of at least 45 participants in each of the two study groups who receive a genomic result to better understand the lived experience of adolescents with an actionable genomic finding and their parents. Data collection will continue after the grant funding ends because of Geisinger Research Division's commitment to following the study cohort. To address the legal specific aim, Dr. Wagner will lead the study team's legal experts in examining and monitoring the loss of chance doctrine in medical malpractice cases in federal and state courts across the United States and in monitoring legislative developments relating to the loss of chance doctrine as it applies to returning adult-onset genomic results to children.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric MyCode participant (ages 0-17) OR
* Parent of a pediatric MyCode participant who has given assent to participate in this study.

Exclusion Criteria:

* Individuals who have already had genetic counseling for any of the actionable target conditions as part of their routine clinical care.
* Individuals who have already had genetic counseling for any of the actionable target conditions through their participation in another research study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) | Baseline, 1, 6, & 12 months post-disclosure
  The HADS questionnaire is a 14-item scale comprised of seven questions for anxiety and seven questions for depression. Each item is scored from 0-3. The total scoring is as follows: 8-10 = Mild, 11-14 = Moderate, 15-21 = Severe. Scoring for anxiety and depression are to be completed separately. For both scales, a total score of less than 7 indicates non-cases.
The General Functioning 12-item subscale (GF12) of The McMaster Family Assessment Device (FAD) | Baseline, 1, 6, & 12 months post-disclosure
  The GF12 subscale is made up of 12 items, six items that reflect healthy family functioning and the other six items reflecting unhealthy functioning. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scale for the negatively worded items reversed.
  The total score is then divided by the number of items on the subscale giving a total score ranging from 1.0 (best functioning) to 4.0 (worse functioning)
Health-Related Quality of Life (HRQOL) | Baseline, 1, 6, & 12 months post-disclosure
  Healthy days are the positive complementary form of unhealthy days. Healthy days estimates the number of recent days when a person's physical and mental health was good (or better) and is calculated by subtracting the number of unhealthy days from 30 days.
  Unhealthy days are an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. To obtain this estimate, responses to questions 2 and 3 are combined to calculate a summary index of overall unhealthy days, with a logical maximum of 30 unhealthy days. For example, a person who reports 4 physically unhealthy days and 2 mentally unhealthy days is assigned a value of 6 unhealthy days, and someone who reports 30 physically unhealthy days and 30 mentally unhealthy days is assigned the maximum of 30 unhealthy days.
Uptake of cascade testing | 12 months post-disclosure to pediatric proband
  Uptake of cascade testing (yes/no) among parents.
Initiation of risk reduction behavior | 12 months post-disclosure to pediatric proband
  Initiation of risk reduction behavior (yes/no) among parents with familial gene variant.

SECONDARY OUTCOMES:
Body Image instrument | Baseline, 1, 6, & 12 months post-disclosure
  Change in adolescents' body image measured using the Body image instrument.
Self-Esteem Scale | Baseline, 1, 6, & 12 months post-disclosure
  The Self-Esteem Scale is made up on 10 items to measure self-esteem. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item.
  The scale can also be scored by totaling the individual 4-point items after reverse-scoring the negatively worded items.
Decision Regret scale | 1 & 12 months post-disclosure
  The Decision Regret Scale is made up of 5 items that address the notion of regret in a variety of ways. Scoring on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scale for the negatively worded items.
  The total score is taken from the mean of the 5 items.
Genetic Counseling Satisfaction Scale (GCSS) | 1 month post-disclosure
  The GCSS is a 6-item Likert scale that assesses participant satisfaction with the process and content of genetic counseling. Scoring on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scale for the negatively worded items.
  The total score is taken from the mean of the 6 items.
Children's Revised Impact of Events scale | 1, 6, &12 months post-disclosure
  The CRIES is a 13-item scale developed as a screening instrument for children at risk of developing PTSD after experiencing a traumatic event. It includes four items measuring intrusion, four items measuring avoidance and five items measuring arousal. Each item is rated on a four-point scale (Not at all, Rarely, Sometimes, Often), scored 0, 1, 3, 5 with no reversed items. The total score indicates the severity of a child's posttraumatic stress reactions with a range from 0 to 65.
  A score of 30 and above has been confirmed as the most effective cut-off score for screening cases of PTSD
Psychological Adaptation to Genetic Information scale (PAGIS) | 1, 6, & 12 months post-disclosure
  This scale consists of both positively and negatively worded statements that are rated on a 1-6 Likert scale (from 1 for strongly disagree to 6 for strongly agree). The respondent's overall health and health of the affected child (where applicable) is assessed using 5-point likert type items.
Health Education Impact Questionnaire (heiQ) | 1, 6, & 12 months post-disclosure
  The Self-Monitoring and Insight scale captures an individuals' ability to monitor their condition, and their physical and or emotional responses that leads to insight and appropriate action/s to self-manage. It is made up of 7 items, scored by summing item responses and dividing by the number of scale items Scoring is done on a 4-point scale (from 1 for strongly disagree to 4 for strongly agree).
  The Health Services Navigation scale aims to capture the positive impact of social engagement and support that evolves through interaction with others and the impact may arise from interaction with others sharing similar health-related life experiences.
  It is made up of 5 items, scored by summing item responses and dividing by the number of scale items Scoring is done on a 4-point scale (from 1 for strongly disagree to 4 for strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Adam H Buchanan, MS, MPH, CGC, Principal Investigator — Geisinger - Department of Genomic Health
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of his/her responsibilities for the proposed study, the Geisinger Data Broker will work under the guidance of Dr. Kirchner to prepare a cleaned, de-identified copy of each quantitative data set used to support each publication that derives from the study. Data will be stripped of identifiers according to the Safe Harbor method of de-identification (https://www.hhs.gov/hipaa/for-professionals/privacy/special-topics/de-identification/index.html).
  These data and related information (participant flow, baseline characteristics, outcome measures and statistical analyses) will then be uploaded to ClinicalTrials.gov within four weeks of acceptance of the corresponding publication. If applicable, the Data Broker will work with the project manager to upload data on adverse events to ClinicalTrials.gov on the same time schedule.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Within four weeks of acceptance of the corresponding publication.

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Boterhoven de Haan KL, Hafekost J, Lawrence D, Sawyer MG, Zubrick SR. Reliability and validity of a short version of the general functioning subscale of the McMaster Family Assessment Device. Fam Process. 2015 Mar;54(1):116-23. doi: 10.1111/famp.12113. Epub 2014 Nov 11. PMID 25385473
- [Background] Moos R, Moos B. Family Environment Scale Manual: Development, Applications, Research. 3rd ed. Palo Alto, CA: Consulting Psychologist Press; 1994
- [Background] Rosenberg M. Society and the adolescent self-image. Princeton, NJ: Princeton University Press; 1965
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] DeMarco TA, Peshkin BN, Mars BD, Tercyak KP. Patient satisfaction with cancer genetic counseling: a psychometric analysis of the Genetic Counseling Satisfaction Scale. J Genet Couns. 2004 Aug;13(4):293-304. doi: 10.1023/b:jogc.0000035523.96133.bc. PMID 19736695
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Patenaude AF, Dorval M, DiGianni LS, Schneider KA, Chittenden A, Garber JE. Sharing BRCA1/2 test results with first-degree relatives: factors predicting who women tell. J Clin Oncol. 2006 Feb 1;24(4):700-6. doi: 10.1200/JCO.2005.01.7541. PMID 16446344
- [Background] Gray SW, Martins Y, Feuerman LZ, Bernhardt BA, Biesecker BB, Christensen KD, Joffe S, Rini C, Veenstra D, McGuire AL; CSER Consortium Outcomes and Measures Working Group. Social and behavioral research in genomic sequencing: approaches from the Clinical Sequencing Exploratory Research Consortium Outcomes and Measures Working Group. Genet Med. 2014 Oct;16(10):727-35. doi: 10.1038/gim.2014.26. Epub 2014 Mar 13. PMID 24625446
- [Background] DuBenske LL, Burke Beckjord E, Hawkins RP, Gustafson DH. Psychometric evaluation of the Health Information Orientation Scale: a brief measure for assessing health information engagement and apprehension. J Health Psychol. 2009 Sep;14(6):721-30. doi: 10.1177/1359105309338892. PMID 19687109
- [Background] Bradbury AR, Patrick-Miller L, Schwartz LA, Egleston BL, Henry-Moss D, Domchek SM, Daly MB, Tuchman L, Moore C, Rauch PK, Shorter R, Karpink K, Sands CB. Psychosocial Adjustment and Perceived Risk Among Adolescent Girls From Families With BRCA1/2 or Breast Cancer History. J Clin Oncol. 2016 Oct 1;34(28):3409-16. doi: 10.1200/JCO.2015.66.3450. Epub 2016 Aug 22. PMID 27551110
- [Background] Lupo PJ, Robinson JO, Diamond PM, Jamal L, Danysh HE, Blumenthal-Barby J, Lehmann LS, Vassy JL, Christensen KD, Green RC, McGuire AL; MedSeq Project team. Patients' perceived utility of whole-genome sequencing for their healthcare: findings from the MedSeq project. Per Med. 2016 Jan 1;13(1):13-20. doi: 10.2217/pme.15.45. Epub 2016 Jan 8. PMID 27019659
- [Background] Schwartz MD, Kaufman E, Peshkin BN, Isaacs C, Hughes C, DeMarco T, Finch C, Lerman C. Bilateral prophylactic oophorectomy and ovarian cancer screening following BRCA1/BRCA2 mutation testing. J Clin Oncol. 2003 Nov 1;21(21):4034-41. doi: 10.1200/JCO.2003.01.088. PMID 14581427
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Kaphingst KA, Facio FM, Cheng MR, Brooks S, Eidem H, Linn A, Biesecker BB, Biesecker LG. Effects of informed consent for individual genome sequencing on relevant knowledge. Clin Genet. 2012 Nov;82(5):408-15. doi: 10.1111/j.1399-0004.2012.01909.x. Epub 2012 Aug 7. PMID 22694298
- [Background] Buchanan AH, Voils CI, Schildkraut JM, Fine C, Horick NK, Marcom PK, Wiggins K, Skinner CS. Adherence to Recommended Risk Management among Unaffected Women with a BRCA Mutation. J Genet Couns. 2017 Feb;26(1):79-92. doi: 10.1007/s10897-016-9981-6. Epub 2016 Jun 6. PMID 27265406
- [Background] Giannopoulou I, Smith P, Ecker C, Strouthos M, Dikaiakou A, Yule W. Factor structure Children's Revised Impact of Events (CRIES) Scale with children exposed to earthquake Pers Individ Diff. 2006;40(5):1027-1037
- [Background] Read CY, Perry DJ, Duffy ME. Design and psychometric evaluation of the Psychological Adaptation to Genetic Information Scale. J Nurs Scholarsh. 2005;37(3):203-8. doi: 10.1111/j.1547-5069.2005.00036.x. PMID 16235859
- [Background] Osborne RH, Elsworth GR, Whitfield K. The Health Education Impact Questionnaire (heiQ): an outcomes and evaluation measure for patient education and self-management interventions for people with chronic conditions. Patient Educ Couns. 2007 May;66(2):192-201. doi: 10.1016/j.pec.2006.12.002. Epub 2007 Feb 22. PMID 17320338
- [Background] McDermott E, Moloney J, Rafter N, Keegan D, Byrne K, Doherty GA, Cullen G, Malone K, Mulcahy HE. The body image scale: a simple and valid tool for assessing body image dissatisfaction in inflammatory bowel disease. Inflamm Bowel Dis. 2014 Feb;20(2):286-90. doi: 10.1097/01.MIB.0000438246.68476.c4. PMID 24374873
- [Background] Greco LA, Lambert W, Baer RA. Psychological inflexibility in childhood and adolescence: development and evaluation of the Avoidance and Fusion Questionnaire for Youth. Psychol Assess. 2008 Jun;20(2):93-102. doi: 10.1037/1040-3590.20.2.93. PMID 18557686
- [Background] CDC. Office of Public Health Genomics - Genomic Tests and Family History by Levels of Evidence.2014; http://www.cdc.gov/genomics/gtesting/tier.htm.
- [Background] Green ED, Guyer MS; National Human Genome Research Institute. Charting a course for genomic medicine from base pairs to bedside. Nature. 2011 Feb 10;470(7333):204-13. doi: 10.1038/nature09764. PMID 21307933
- [Derived] Savatt JM, Urban GM, Floyd AE, Leitzel T, Murray JAC, Hu Y, Williams MS, Buchanan AH. Performance of recommended management among pediatric patients identified through genomic screening. Transl Behav Med. 2025 Jan 16;15(1):ibaf065. doi: 10.1093/tbm/ibaf065. PMID 41193187
- [Derived] Savatt JM, Wagner JK, Joffe S, Rahm AK, Williams MS, Bradbury AR, Davis FD, Hergenrather J, Hu Y, Kelly MA, Kirchner HL, Meyer MN, Mozersky J, O'Dell SM, Pervola J, Seeley A, Sturm AC, Buchanan AH. Pediatric reporting of genomic results study (PROGRESS): a mixed-methods, longitudinal, observational cohort study protocol to explore disclosure of actionable adult- and pediatric-onset genomic variants to minors and their parents. BMC Pediatr. 2020 May 15;20(1):222. doi: 10.1186/s12887-020-02070-4. PMID 32414353

DOCUMENTS (1):
  • Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT03832985/ICF_000.pdf